CLINICAL TRIAL: NCT01298895
Title: Optical Low Coherence Reflectometry Enables Preoperative Detection of Zonular Weakness in Pseudoexfoliation Syndrome
Status: Completed | Type: Observational
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Damir Bosnar, PhD, Eye Clinic, General hospital Sveti Duh, Zagreb, Croatia
Other Study IDs: 0192/09.01.2009.
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2009-01

CONDITIONS: Pseudoexfoliation Syndrome
Keywords: optical components; pseudoexfoliation; cataract; LENSTAR® LS 900®
MeSH Terms: conditions — Exfoliation Syndrome; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PEX group: The first group consisted of 47 eyes with cataract complicated with pseudoexfoliation syndrome (PEX).
- control group: The control group included 177 eyes with uncomplicated cataract in eyes without other ocular pathology

SUMMARY:
The purpose of the study was to evaluate optical ocular components in patients with pseudoexfoliation syndrome using optical low coherence reflectometry. A prospective cohort study of 224 eyes of patients planned for cataract surgery was conducted from January 2009 until July 2009. Patients were divided in two groups: the first group of 47 eyes with cataract complicated with pseudoexfoliation syndrome and the control group of 177 eyes with uncomplicated cataract. Each group was further divided into two subgroups based on its refractive state: emmetropes and hypermetropes. The optical low coherence reflectometry biometer LENSTAR® LS 900® was used to define ocular optical components.

DETAILED DESCRIPTION:
Material and methods A prospective cohort study of 224 eyes of patients planned for cataract surgery was conducted at the University Eye Clinic, General Hospital Sveti Duh, Zagreb, Croatia. The inclusion criteria was age of patients over 40 years. Sex and refractive eye state were randomly chosen out of all cataract patients operated at the Clinic from January 2009 until July 2009. Patients were divided in two groups. The first group consisted of 47 eyes with cataract complicated with PEX. The control group included 177 eyes with uncomplicated cataract in eyes without other ocular pathology. Refractive state was defined by preoperatively calculated emmetropisation intraocular lens (IOL) value done by LENSTAR LS 900®. Emmetropes had IOL value of 20-22 diopters and hypermetropes of more than 22 diopters. There were no myopic patients defined as IOL value less than 20 diopters in the PEX group operated at the Clinic in the defined time. Consequently, there were no myopic patients included in the control group. The PEX group and the control group were further divided into two subgroups: emmetropes and hypermetropes. LENSTAR LS 900® was used to measure ocular optical components 3-9: axial length (AL), central corneal thickness (CCT), anterior chamber depth (ACD), lens thickness (LT), retinal thickness (RT), keratometry values (keratometry of the steepest meridian (K1), keratometry of the flattest meridian (K2), its position regarding horizontal line (AXIS) and the difference between K1 and K2 (astigmatism, AST), horizontal diameter of iris (WTW) and pupillary diameter (PD). Ethics committee approval of General Hospital Sveti Duh, Zagreb, Croatia, was secured for the study reported. All study procedures adhered to the recommendations of the Declaration of Helsinki. Written consent was obtained from all patients prior to their inclusion in the study. Sample size was defined in a way to provide sufficient statistical power of the study, which was in this case over 90%. Descriptive statistics and Student's t-test were used for data evaluation. Value of p<0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* age of patients over 40 years old
* must have cataract
* for the PEX group must have cataract complicated with PEX

Exclusion criteria:

* age below 40 years old
* absence of cataract
* presence of other ocular pathology in the control group

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort study of 224 eyes of patients planned for cataract surgery was conducted at the University Eye Clinic, General hospital Sveti Duh, Zagreb, Croatia. The inclusion criteria was age of patients over 40 years. Sex and refractive eye state were randomly chosen out of all cataract patients operated at the Clinic from January 2009 until July 2009.
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mladen Bušić, Assoc.Prof., Study Director — University Eye Clinic, General hospital Sveti Duh, Zagreb, Croatia
Locations (1):
- General Hospital Sveti Duh, Zagreb, Croatia

REFERENCES:
- [Background] Busic M, Kastelan S. Pseudoexfoliation syndrome and cataract surgery by phacoemulsification. Coll Antropol. 2005;29 Suppl 1:163-6. PMID 16193703
- [Background] Scorolli L, Scorolli L, Campos EC, Bassein L, Meduri RA. Pseudoexfoliation syndrome: a cohort study on intraoperative complications in cataract surgery. Ophthalmologica. 1998;212(4):278-80. doi: 10.1159/000027307. PMID 9672219
- [Background] Buckhurst PJ, Wolffsohn JS, Shah S, Naroo SA, Davies LN, Berrow EJ. A new optical low coherence reflectometry device for ocular biometry in cataract patients. Br J Ophthalmol. 2009 Jul;93(7):949-53. doi: 10.1136/bjo.2008.156554. Epub 2009 Apr 19. PMID 19380310
- [Background] Cruysberg LP, Doors M, Verbakel F, Berendschot TT, De Brabander J, Nuijts RM. Evaluation of the Lenstar LS 900 non-contact biometer. Br J Ophthalmol. 2010 Jan;94(1):106-10. doi: 10.1136/bjo.2009.161729. Epub 2009 Aug 18. PMID 19692383
- [Background] Rohrer K, Frueh BE, Walti R, Clemetson IA, Tappeiner C, Goldblum D. Comparison and evaluation of ocular biometry using a new noncontact optical low-coherence reflectometer. Ophthalmology. 2009 Nov;116(11):2087-92. doi: 10.1016/j.ophtha.2009.04.019. Epub 2009 Sep 10. PMID 19744720
- [Background] Hoffer KJ, Shammas HJ, Savini G. Comparison of 2 laser instruments for measuring axial length. J Cataract Refract Surg. 2010 Apr;36(4):644-8. doi: 10.1016/j.jcrs.2009.11.007. PMID 20362858
- [Background] Liampa Z, Kynigopoulos M, Pallas G, Gerding H. Comparison of two partial coherence interferometry devices for ocular biometry. Klin Monbl Augenheilkd. 2010 Apr;227(4):285-8. doi: 10.1055/s-0029-1245182. Epub 2010 Apr 20. PMID 20408075
- [Background] Bjelos Roncevic M, Busic M, Cima I, Kuzmanovic Elabjer B, Bosnar D, Miletic D. Comparison of optical low-coherence reflectometry and applanation ultrasound biometry on intraocular lens power calculation. Graefes Arch Clin Exp Ophthalmol. 2011 Jan;249(1):69-75. doi: 10.1007/s00417-010-1509-4. Epub 2010 Sep 18. PMID 20853004
- [Background] Bjelos Roncevic M, Busic M, Cima I, Kuzmanovic Elabjer B, Bosnar D, Miletic D. Intraobserver and interobserver repeatability of ocular components measurement in cataract eyes using a new optical low coherence reflectometer. Graefes Arch Clin Exp Ophthalmol. 2011 Jan;249(1):83-7. doi: 10.1007/s00417-010-1546-z. Epub 2010 Oct 28. PMID 20981435
- [Background] Karger RA, Jeng SM, Johnson DH, Hodge DO, Good MS. Estimated incidence of pseudoexfoliation syndrome and pseudoexfoliation glaucoma in Olmsted County, Minnesota. J Glaucoma. 2003 Jun;12(3):193-7. doi: 10.1097/00061198-200306000-00002. PMID 12782834
- [Background] Klein BE, Klein R, Lee KE. Incidence of age-related cataract over a 10-year interval: the Beaver Dam Eye Study. Ophthalmology. 2002 Nov;109(11):2052-7. doi: 10.1016/s0161-6420(02)01249-6. PMID 12414414
- [Background] Mccarty CA, Taylor HR. Pseudoexfoliation syndrome in Australian adults. Am J Ophthalmol. 2000 May;129(5):629-33. doi: 10.1016/s0002-9394(99)00466-3. PMID 10844055
- [Background] Bayramlar H, Ozden S, Ergin M, Tutarli H. Ultrasonografic measurement of ocular refractive components in eyes with various refractive states. T Klin Oftalmoloji 3:90-94, 1994.
- [Background] Bartholomew RS. Anterior chamber depth in eyes with pseudoexfoliation. Br J Ophthalmol. 1980 May;64(5):322-3. doi: 10.1136/bjo.64.5.322. PMID 7437392
- [Background] Kuchle M, Viestenz A, Martus P, Handel A, Junemann A, Naumann GO. Anterior chamber depth and complications during cataract surgery in eyes with pseudoexfoliation syndrome. Am J Ophthalmol. 2000 Mar;129(3):281-5. doi: 10.1016/s0002-9394(99)00365-7. PMID 10704540
- [Background] Jünemann A, Martus P, Händel A, Naumann GOH. Ocular dimensions in pseudoexfoliation syndrome. Ophthalmic Res 29:88, 1997.
- [Background] Kaneda J, Sasaki H, Nagai K, Fujisawa A, Kawakami Y, Sakamoto A, N Takahashi N, Sasaki K. Forward Malposition of the Crystalline Lens in Pseudoexfoliation Syndrome. Invest Ophthalmol Vis Sci 43, 2002.
- [Background] Lanzl IM, Merte RL, Graham AD. Does head positioning influence anterior chamber depth in pseudoexfoliation syndrome? J Glaucoma. 2000 Jun;9(3):214-8. doi: 10.1097/00061198-200006000-00003. PMID 10877371
- [Background] Arnarsson A, Damji KF, Sverrisson T, Sasaki H, Jonasson F. Pseudoexfoliation in the Reykjavik Eye Study: prevalence and related ophthalmological variables. Acta Ophthalmol Scand. 2007 Dec;85(8):822-7. doi: 10.1111/j.1600-0420.2007.01051.x. PMID 18028119
- [Background] Salzmann M. The Anatomy and Histology of the Human Eyeball , trans. E. V. L. Brown. University of Chicago Press, Chicago, 1912.
- [Background] Suzuki R, Kurimoto S. Intraocular muscle function in pseudoexfoliation syndrome. Ophthalmologica. 1992;204(4):192-8. doi: 10.1159/000310293. PMID 1513550
- [Background] Naseem A. Cataract surgery in patients with pseudoexfoliation. [Dissertation]. Karachi: College of Physicians & Surgeons :111, 2002.
- [Background] Yulek F, Konukseven OO, Cakmak HB, Orhan N, Simsek S, Kutluhan A. Comparison of the pupillometry during videonystagmography in asymmetric pseudoexfoliation patients. Curr Eye Res. 2008 Mar;33(3):263-7. doi: 10.1080/02713680801915284. PMID 18350437
- [Background] Repo LP, Naukkarinen A, Paljarvi L, Terasvirta ME. Pseudoexfoliation syndrome with poorly dilating pupil: a light and electron microscopic study of the sphincter area. Graefes Arch Clin Exp Ophthalmol. 1996 Mar;234(3):171-6. doi: 10.1007/BF00462029. PMID 8720716
- [Background] Prince AM, Ritch R. Clinical signs of the pseudoexfoliation syndrome. Ophthalmology. 1986 Jun;93(6):803-7. doi: 10.1016/s0161-6420(86)33664-9. PMID 3737125
- [Background] Mohamed NY, Hassan MN, Ali NA, Binnawi KH. Central Corneal Thickness in Sudanese Population. Sud J Ophthalmol 1:29-32, 2009.
- [Background] Oliveira C, Tello C, Liebmann J, Ritch R. Central corneal thickness is not related to anterior scleral thickness or axial length. J Glaucoma. 2006 Jun;15(3):190-4. doi: 10.1097/01.ijg.0000212220.42675.c5. PMID 16778639
- [Background] Chen MJ, Liu YT, Tsai CC, Chen YC, Chou CK, Lee SM. Relationship between central corneal thickness, refractive error, corneal curvature, anterior chamber depth and axial length. J Chin Med Assoc. 2009 Mar;72(3):133-7. doi: 10.1016/S1726-4901(09)70038-3. PMID 19299220
- [Background] Hepsen IF, Yagci R, Keskin U. Corneal curvature and central corneal thickness in eyes with pseudoexfoliation syndrome. Can J Ophthalmol. 2007 Oct;42(5):677-80. doi: 10.3129/i07-145. PMID 17891195
- [Background] Shah S, Chatterjee A, Mathai M, Kelly SP, Kwartz J, Henson D, McLeod D. Relationship between corneal thickness and measured intraocular pressure in a general ophthalmology clinic. Ophthalmology. 1999 Nov;106(11):2154-60. doi: 10.1016/S0161-6420(99)90498-0. PMID 10571352
- [Background] Ganguli D, Roy IS, Biswas SK, Sengupta M. Study of corneal power and diameter in simple refractive error. Indian J Ophthalmol. 1975 Apr;23(1):6-11. No abstract available. PMID 1158423